CLINICAL TRIAL: NCT05043142
Title: Exhaustive, Cross-sectional, Non-interventional, Multicenter Retrospective Epidemiological Study of the COVID-2019 Incidence and Prevention Methods of SARS, Including COVID-2019, Among Staff of Participating Organizations.
Brief Title: Epidemiological Study of the COVID-2019 in Participating Organizations.
Status: Completed | Type: Observational
Sponsor: Yuria-Pharm (Industry)
Collaborators: Pharmaxi LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: EpidProtect-21
Record Dates: First submitted 2021-09-10; First posted 2021-09-14 (Actual); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Prevention; prophylactics; incidence; severity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ELISA test for the antibodies to COVID-2019. — Each subject will be assigned an individual number, which will be used for conduction of a rapid ELISA test for the antibodies to COVID-2019. Subjects will be notified of the test results.

SUMMARY:
Exhaustive, cross-sectional, non-interventional, multicenter retrospective epidemiological study, case study aimed to determine the relationship between the systematic use of prophylactics to prevent SARS, including COVID-2019, and the risks of incidence and serious complications of COVID-2019 among staff of participating organizations.

DETAILED DESCRIPTION:
Coronaviruses are a large family of viruses that might cause illness in animals or humans. SARS-CoV-2 is an enveloped, single-stranded RNA virus of the β genus. It can cause respiratory illness named COVID-19, the severity of which varies from asymptomatic to severe, and which can lead to the patient's death of the long-term consequences (so-called post-COVID syndrome). The virus has spread globally and been declared a Public Health Emergency of International Concern by WHO in January 30, 2020.

The first case of COVID-19 in Ukraine was detected in early March, 2020. 1273475 cases of the disease have been registered in Ukraine as at February 15, 2021.

Quarantine restrictions and other anti-epidemic measures established in Ukraine and their results are the subject of wide debate.

Own anti-epidemic measures, in addition to those established by the Government, have also been implemented by numerous representatives of the public sector, non-governmental organizations and business.

The company management of the participating organizations decided to provide their staff with prophylactic tools and recommendations for COVID-19 prevention.

The study aims to identify the incidence, characteristics of cases and their relationship with the preventive measures used.

Each subject will be assigned an individual number, which will be used for conduction of a rapid ELISA test for the antibodies to COVID-2019. Subjects will be notified of the test results.

The questionnaires will be conducted when the subject enters the data in the electronic case report form after signing the consent to processing of personal data.

For the purposes of analysis, the subject enters his individual number in the questionnaire, as well as number of a rapid ELISA test for antibodies to COVID-2019 and its result. The entered data will be compared with the databases which contain the results of rapid ELISA tests.

The questionnaire includes questions related to the main risks and protective factors of the COVID-2019 disease: demographic, anthropometric data, lifestyle data, prophylactics methods, subject's costs spent on COVID-2019 prophylactics.

For subjects who had the COVID-2019 case, a separate block of questionnaire was created to collect data on prophylactics, treatment of COVID-2019, the course of the disease and the consequences of the disease case, as well as costs spent on COVID-2019 treatment.

The completeness of entered data in the electronic case report form will be controlled by specially designated authorized persons in each participating organization, who were designated by the person responsible for conducting the study in each participating organization.

The correctness of entered data in the electronic case report form will be controlled by remote monitoring.

The questionnaire cannot be completed until all required fields of the case report form have been completed.

A structured description of the available medical documentation for fatal cases of COVID-2019 will be conducted separately.

Demographic, anthropometric data, lifestyle data, prophylactics methods, treatment of COVID-2019, the course of the COVID-2019 case will be described.

Calculation of sample size is not applicable as it is exhaustive study. Participating organizations undertake to organize the involvement in the study of at least 95% of persons employed by participating organizations.

In the context of this data analysis, all the main steps from the primary data to the results of the study will be described separately in the Statistical Analysis Plan.

This study is not intended to accept or reject pre-defined hypotheses, thus statistical analysis will mainly be descriptive.

All types of analysis will be done for the entire available study population with available data.

If there is a sufficient amount of data in the subpopulations, a separate statistical analysis will be performed.

No conditional calculation methods will be applied to the missed values. The statistical generalization will consist of frequency tables of categorical variables (number, %).

For metric variables, descriptive statistics (number of subjects with available observations, number of missed values, mean, standard deviation, median, 25th and 75th percentiles, minimum and maximum) will be presented in tabular form.

Statistical conclusions will be used to assess the potential relationship between the identified variables and the incidence / severity of COVID-2019.

The relationship between the subject's characteristics and the variables of interest will be assessed using a one-dimensional and multidimensional (polynomial) logistic regression model for variables, which have no more than 20% omitted data.

The final model will be selected with a view to minimizing the Akaike information criterion value.

2×2 tables, χ-square were used for calculations of odds ratios. Rough odds ratios and adjusted odds ratios with corresponding 95% confidence intervals and p-values will be generated and presented for both one-dimensional and multidimensional logistics models.

ELIGIBILITY:
Inclusion Criteria:

1. The subject gave the consent to participate in the study and signed the consent to processing of personal data.
2. The subject aged 18 years and older.
3. The subject is employed by one of the participating organizations.

Exclusion Criteria:

The subject may not be included in the study due to non-compliance with the inclusion criteria or due to force majeure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons who are employed by one of the participating organizations (SI National Institute of Phthisiology and Pulmonology named after F.G. Yanovsky; Yuria-Pharm LLC; Infuzia PJSC; Institute Hyalual LLC; Medical Center M.T.K. LLC; InterChem SLC; Diatom LLC).
Sampling Method: Non-Probability Sample
Enrollment: 3632 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tetiana Sprynsian, Study Director — Yuria-Pharm
Locations (7):
- Ukraine (7):
  - SI National Institute of Phthisiology and Pulmonology named after F.G. Yanovsky, Kyiv
  - Institute Hyalual LLC, Kyiv
  - Yuria-Pharm LLC, Kyiv
  - Medical Center M.T.K. LLC, Kyiv
  - Infuzia PJSC, Kyiv
  - Diatom LLC, Kyiv
  - InterChem SLC, Odesa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Ann Bowling. Research Methods in Health: Investigating Health and Health Services, Fourth edition, 2014, Maidenhead, GB. McGraw Hill; Open University Press, 536pp — https://eprints.soton.ac.uk/371922/
- See also: Bernard Rosner. Fundamentals of Biostatistics, Seventh Edition, 2010. — https://www.worldcat.org/title/fundamentals-of-biostatistics/oclc/660057729
- See also: Ann Aschengrau. Essentials of Epidemiology in Public Health, Fourth Edition — https://www.jblearning.com/catalog/productdetails/9781284128352
- See also: Bonita, Ruth, Beaglehole, Robert, Kjellström, Tord & World Health Organization. (2006). Basic epidemiology, 2nd ed. World Health Organization — https://apps.who.int/iris/handle/10665/43541
- See also: Earl Babbie. The Practice of Social Research, Twelfth edition, 2009 — https://www.amazon.com/Earl-R-Babbie-Practice-Research/dp/B004HMCISY

RESULTS

PARTICIPANT FLOW:
Groups:
- Cross-sectional Study on COVID-19: One group study included subjects who employed by one of the following organizations:
  * SI National Institute of Phthisiology and Pulmonology named after F.G. Yanovsky.
  * Yuria-Pharm LLC.
  * Infuzia PJSC.
  * Institute Hyalual LLC.
  * Medical Center M.T.K. LLC.
  * InterChem SLC.
  * Diatom LLC.
Period: Overall Study
Arm/Group | Cross-sectional Study on COVID-19
Started | 3632
Completed | 3443
Not Completed | 189

BASELINE CHARACTERISTICS:
Groups:
- Group One: One group study
Arm/Group | Group One
Number analyzed (Participants) | 3443
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.62 (11.954)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1978
  Male | 1465
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ukraine | 3443
Weight [Mean (Standard Deviation); unit: kg] | 75.97 (16.374)
Height [Mean (Standard Deviation); unit: cm] | 171.11 (9.140)
Number of people in the household [Mean (Standard Deviation); unit: person] | 2.88 (1.250)
Blood group [Count of Participants; unit: Participants]
  I (Type O) | 935
  II (Type A) | 1231
  III (Type B) | 607
  IV (Type AB) | 290
  Not known | 380
Presence of bad habits [Count of Participants; unit: Participants]
  Present | 973
  Absent | 2470
Tobacco smoking / use of other nicotine products [Count of Participants; unit: Participants] | 875
Alcohol consumption [Count of Participants; unit: Participants] | 343
Frequency of alcohol consumption [Count of Participants; unit: Participants]
  Almost everyday (more than 4 tomes a week) | 8
  Rarely (less than 2 times a week) | 301
  Often (more than 2 times a week) | 28
  Everyday | 6
  No | 3100
Other bad habits [Count of Participants; unit: Participants] — Other bad habits were reported by participants if they percieve their behavior as potentially hazardous for thier physical/mental health.
  Participants | 12
Physical activity [Count of Participants; unit: Participants]
  very active (intense physical activity 6-7 days a week) | 394
  slightly active (easy exercises 1-3 times a week) | 1357
  sedentary (easy / no exercise, sedentary work) | 431
  extremely active (intense physical activity everyday) | 107
  moderately active (training / sports 3-5 times a week) | 1154
Changes in diet from March 2020 [Count of Participants; unit: Participants] — This includes all changes in eating habits like exclusion of some nutritional components, consumption of any supplements, regiment or volume of food intake.
  Participants | 234
Chronic diseases [Count of Participants; unit: Participants] — Chronic diseases are defined broadly as conditions that last 1 year or more and require ongoing medical attention or limit activities of daily living or both.
  Participants | 694
Chronic non-infectious diseases [Count of Participants; unit: Participants] | 498
Chronic non-infectious diseases [Count of Participants; unit: Participants]
  bronchial asthma | 29
  coronary heart disease | 42
  hypertensive disease | 180
  COPD (chronic obstructive pulmonary disease) | 19
  tumors (malignant / benign) | 24
  diabetes | 43
  other | 277
  No chronic non-infectious diseases | 2945
Type of diabetes [Count of Participants; unit: Participants]
  I | 9
  II | 34
  No diabetes | 3400
Compensation for chronic non-infectious diseases [Count of Participants; unit: Participants] — Controll over the chronic disease means that participants can manage daily symptoms that affect their quality of life, and avoid acute health problems and complications that can shorten their life expectancy.
  Participants | 253
Systematic treatment of non-infectious diseases [Count of Participants; unit: Participants] | 345
Number of drugs systematically taken for treatment of non-infectious diseases [Count of Participants; unit: Participants]
  1 | 133
  2 | 118
  3 | 45
  4 | 23
  5 | 17
  6 | 3
  7 | 6
  No drugs taken for treatment of of non-infectious diseases | 3098
Chronic infectious diseases [Count of Participants; unit: Participants] — Chronic diseases are defined broadly as conditions caused by the infectious agent (e.g., bacteria, virus, parasite) that last 1 year or more and require ongoing medical attention or limit activities of daily living or both
  Participants | 26
Systematic treatment of infectious diseases [Count of Participants; unit: Participants] | 8
Number of drugs systematically taken for treatment of infectious diseases [Count of Participants; unit: Participants]
  1 | 3
  2 | 3
  3 | 2
  No drugs taken for treatment of infectious diseases | 3435
Frequency of acute respiratory infectious diseases [Count of Participants; unit: Participants]
  1-2 times a year | 1673
  3-4 times a year | 234
  less than 1 time a year | 1495
  more than 4 times a year | 41

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of COVID-2019 Cases.
Description: The incidence of COVID-2019 cases in participating organizations by which study subjects are employed (SI National Institute of Phthisiology and Pulmonology named after F.G. Yanovsky; Yuria-Pharm LLC; Infuzia PJSC; Institute Hyalual LLC; Medical Center M.T.K. LLC; InterChem SLC; Diatom LLC).
  .
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number; unit: COVID-2019 cases per 1000 person
Arm/Group | Group One
Number analyzed (Participants) | 3443
COVID-2019 cases per 1000 person | 259.95

2. Secondary Outcome: The Severity of the COVID-2019 Cases in Participating Organizations.
Description: The severity of the COVID-2019 cases in participating organizations by which study subjects are employed (SI National Institute of Phthisiology and Pulmonology named after F.G. Yanovsky; Yuria-Pharm LLC; Infuzia PJSC; Institute Hyalual LLC; Medical Center M.T.K. LLC; InterChem SLC; Diatom LLC).
Time Frame: 1 visit from March 2021 till June 2021
Measure: Count of Participants; unit: Participants
Arm/Group | Group One
Number analyzed (Participants) | 3443
Participants
  Asymptomatic | 55
  Very severe | 6
  Mild | 451
  Moderate | 315
  Severe | 65
  No COVID Case | 2551

3. Secondary Outcome: Prevention Methods of SARS, Including COVID-2019, Which Were Used by Subject That Had at Least One COVID-2019 Case.
Description: Prevention methods of SARS, including COVID-2019, which were used by subject that had at least one COVID-2019 case. The number of participants is reported for every prevention method separately.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Count of Participants; unit: Participants
Arm/Group | Group One
Number analyzed (Participants) | 878
Participants
  Inhalation antiseptics | 79
  Inhalation antiviral drugs | 60
  Oral systemic antiviral drugs | 124
  Injectable systemic antiviral drugs | 1
  Immunomodulatory drugs | 97
  Vitamins | 140
  Antibiotics | 3
  Herbal drugs | 14
  Homeopathic drugs | 4
  Other drugs | 10
  No Prevention | 346

4. Secondary Outcome: Prevention Methods of SARS, Including COVID-2019, Which Were Used by Subject That Did Not Have Any COVID-2019 Case.
Description: Prevention methods of SARS, including COVID-2019, which were used by subject that did not have any COVID-2019 case. The number of participants is reported for every prevention method separately.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Count of Participants; unit: Participants
Arm/Group | Group One
Number analyzed (Participants) | 842
Participants
  Inhalation antiseptics | 353
  Inhalation antiviral drugs | 366
  Oral systemic antiviral drugs | 583
  Injectable systemic antiviral drugs | 4
  Immunomodulatory drugs | 566
  Vitamins | 523
  Antibiotics | 25
  Herbal drugs | 35
  Homeopathic drugs | 31
  Other drugs | 111

5. Secondary Outcome: Relationship Between the Used Prevention Methods and and the Risk to Have at Least One Case of COVID-2019 Among Staff of Participating Organizations.
Description: Relationship between the used prevention methods and iand the Risk to Have at Least One Case of COVID-2019. among staff of participating organizations.Prevention methods within this outcome includes all prevention methods which were used by subjects. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.875 [0.776 to 0.986]

6. Secondary Outcome: Relationship Between the Presence of Comorbidities, Such as Bronchial Asthma and COPD (Chronic Obstructive Pulmonary Disease), and the Risk to Have at Least One Case of COVID-2019.
Description: Relationship between the presence of comorbidities, such as bronchial asthma and COPD (Chronic obstructive pulmonary disease), and the risk to have at least one case of COVID-2019. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.892 [0.389 to 2.046]

7. Secondary Outcome: Relationship Between the COVID-2019 Case and the Risk of Change of the Course of Comorbidities, Such as Bronchial Asthma and сhronic Obstructive Pulmonary Disease (COPD).
Description: Relationship between the COVID-2019 case and the risk of change of the course of comorbidities, such as bronchial asthma and сhronic obstructive pulmonary disease (COPD). Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.523 [0.300 to 0.911]

8. Secondary Outcome: Relationship Between Different Strategies and Combinations of Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between different strategies and combinations of drugs used for prophylactics at any time from March 2020 and the risk of having a COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.949 [0.911 to 0.989]

9. Secondary Outcome: Relationship Between Different Strategies and Combinations of Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a Severe COVID-2019 Case.
Description: Relationship between different strategies and combinations of drugs used for prophylactics at any time from March 2020 and the risk of having a severe COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 1.002 [0.958 to 1.047]

10. Secondary Outcome: Relationship Between Different Strategies and Combinations of Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between different strategies and combinations of drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.981 [0.948 to 1.014]

11. Post Hoc Outcome: Relationship Between Inhalation Antiseptics + Oral Systemic Antiviral Drugs + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between inhalation antiseptics + oral systemic antiviral drugs + other drugs used for prophylactics at any time from March 2020 and the risk of having a COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.744 [0.729 to 0.759]

12. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Immunomodulatory Drugs + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + immunomodulatory drugs + other drugs used for prophylactics at any time from March 2020 and the risk of having a COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.743 [0.728 to 0.758]

13. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Oral Systemic Antiviral Drugs + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + oral systemic antiviral drugs + other drugs used for prophylactics at any time from March 2020 and the risk of having a COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.744 [0.729 to 0.759]

14. Post Hoc Outcome: Relationship Between Oral Systemic Antiviral Drugs + Vitamins + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between oral systemic antiviral drugs + vitamins + other drugs used for prophylactics at any time from March 2020 and the risk of having a COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.742 [0.727 to 0.757]

15. Post Hoc Outcome: Relationship Between Specific Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between specific prophylactics at any time from March 2020 and the risk of having a COVID-2019 case.
  Specific prophylactics included inhalation antiseptics, inhalation antiviral drugs, oral systemic antiviral drugs, injectable systemic antiviral drugs, immunomodulatory drugs and antibiotics.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 1.013 [0.949 to 1.082]

16. Post Hoc Outcome: Relationship Between Nonspecific Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between nonspecific prophylactics at any time from March 2020 and the risk of having a COVID-2019 case.
  Nonspecific prophylactics included vitamins, herbal drugs, homeopathic drugs and other drugs.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 11.291 [2.959 to 43.078]

17. Post Hoc Outcome: Relationship Between Combined Prophylactics at Any Time From March 2020 and the Risk of Having a COVID-2019 Case.
Description: Relationship between combined prophylactics at any time from March 2020 and the risk of having a COVID-2019 case.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.877 [0.841 to 0.914]

18. Post Hoc Outcome: Relationship Between Inhalation Antiseptics + Oral Systemic Antiviral Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a Severe COVID-2019 Case.
Description: Relationship between inhalation antiseptics + oral systemic antiviral drugs used for prophylactics at any time from March 2020 and the risk of having a severe COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.918 [0.9 to 0.937]

19. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Oral Systemic Antiviral Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Having a Severe COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + oral systemic antiviral drugs used for prophylactics at any time from March 2020 and the risk of having a severe COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.918 [0.9 to 0.937]

20. Post Hoc Outcome: Relationship Between Nonspecific Prophylactics at Any Time From March 2020 and the Risk of Having a Severe COVID-2019 Case.
Description: Relationship between nonspecific prophylactics at any time from March 2020 and the risk of having a severe COVID-2019 case.
  Nonspecific prophylactics included vitamins, herbal drugs, homeopathic drugs and other drugs.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.953 [0.885 to 1.026]

21. Post Hoc Outcome: Relationship Between Specific Prophylactics at Any Time From March 2020 and the Risk of Having a Severe COVID-2019 Case.
Description: Relationship between specific prophylactics at any time from March 2020 and the risk of having a severe COVID-2019 case.
  Specific prophylactics included inhalation antiseptics, inhalation antiviral drugs, oral systemic antiviral drugs, injectable systemic antiviral drugs, immunomodulatory drugs and antibiotics.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.995 [0.935 to 1.059]

22. Post Hoc Outcome: Relationship Between Combined Prophylactics at Any Time From March 2020 and the Risk of Having a Severe COVID-2019 Case.
Description: Relationship between combined prophylactics at any time from March 2020 and the risk of having a severe COVID-2019 case.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: RR
Arm/Group | Group One
Number analyzed (Participants) | 3443
RR | 1.026 [0.961 to 1.095]

23. Post Hoc Outcome: Relationship Between Vitamins + Herbal Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between vitamins + herbal drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

24. Post Hoc Outcome: Relationship Between Vitamins + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between vitamins + other drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

25. Post Hoc Outcome: Relationship Between Inhalation Antiseptics + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiseptics + other drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

26. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + other drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

27. Post Hoc Outcome: Relationship Between Oral Systemic Antiviral Drugs + Herbal Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between oral systemic antiviral drugs + herbal drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

28. Post Hoc Outcome: Relationship Between Immunomodulatory Drugs + Herbal Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between immunomodulatory drugs + herbal drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

29. Post Hoc Outcome: Relationship Between Inhalation Antiseptics + Oral Systemic Antiviral Drugs + Vitamins Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiseptics + oral systemic antiviral drugs + vitamins used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.927 to 0.959]

30. Post Hoc Outcome: Relationship Between Inhalation Antiseptics + Immunomodulatory Drugs + Vitamins Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiseptics + immunomodulatory drugs + vitamins used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

31. Post Hoc Outcome: Relationship Between Inhalation Antiseptics + Vitamins + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiseptics + vitamins + other drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

32. Post Hoc Outcome: Relationship Between Immunomodulatory Drugs + Vitamins + Herbal Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between immunomodulatory drugs + vitamins + herbal drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

33. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Oral Systemic Antiviral Drugs + Vitamins Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + oral systemic antiviral drugs + vitamins used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.927 to 0.959]

34. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Immunomodulatory Drugs + Vitamins Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + immunomodulatory drugs + vitamins used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

35. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Vitamins + Other Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + vitamins + other drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

36. Post Hoc Outcome: Relationship Between Inhalation Antiviral Drugs + Vitamins + Herbal Drugs Used for Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between inhalation antiviral drugs + vitamins + herbal drugs used for prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.943 [0.928 to 0.959]

37. Post Hoc Outcome: Relationship Between Specific Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between specific prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case.
  Specific prophylactics included inhalation antiseptics, inhalation antiviral drugs, oral systemic antiviral drugs, injectable systemic antiviral drugs, immunomodulatory drugs and antibiotics. Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.998 [0.947 to 1.051]

38. Post Hoc Outcome: Relationship Between Nonspecific Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between nonspecific prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case.
  Nonspecific prophylactics included vitamins, herbal drugs, homeopathic drugs and other drugs.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.978 [0.909 to 1.052]

39. Post Hoc Outcome: Relationship Between Combined Prophylactics at Any Time From March 2020 and the Risk of Hospitalization of Persons Who Had at Least One COVID-2019 Case.
Description: Relationship between combined prophylactics at any time from March 2020 and the risk of hospitalization of persons who had at least one COVID-2019 case.
  Measure of outcome is risk ratio (RR), also called relative risk, compares the risk of a health event (disease, injury, risk factor, or death) among one group with the risk among another group. It does so by dividing the risk (incidence proportion, attack rate) in group 1 by the risk (incidence proportion, attack rate) in group 2. If the risk ratio is 1 (or close to 1), it suggests no difference or little difference in risk (incidence in each group is the same). A risk ratio > 1 suggests an increased risk of that outcome in the exposed group. A risk ratio < 1 suggests a reduced risk in the exposed group.
Time Frame: 1 visit from March 2021 till June 2021
Measure: Number (95% Confidence Interval); unit: Risk Ratio
Arm/Group | Group One
Number analyzed (Participants) | 3443
Risk Ratio | 0.976 [0.937 to 1.017]

ADVERSE EVENTS:
Time Frame: No data on adverse events were collected.
Description: The number of participants at risk for Serious Adverse Events, All-Cause Mortality, Other (Not Including Serious) Adverse Events is zero, because this is observational retrospective study.
Arm/Group | Group One
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
* Probable selection bias (employed, but not present at office).
* Long-term data collection there is a difference in the duration of action of the exposure factor.
* The retrospective study design has limitations on the completeness and accuracy of the data provided by the study subjects.
* The direction of the relationship cannot be determined for all relationships (there may be an inverse relationship).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT05043142/Prot_SAP_000.pdf